CLINICAL TRIAL: NCT06545019
Title: Study of Informative Video On Alleviating Perioperative Anxiety And Improving Satisfaction Score In Obstetric Patient Undergoing Elective Lower Segment Caesarean Section Under Spinal Anaesthesia
Brief Title: Informative Video to Alleviate Anxiety and Improve Satisfaction in Elective Caesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Hadri Kamarrudin, Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202459-13718
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pre-operative Anxiety; Spinal Anesthesia; Satisfaction, Patient
Keywords: Informative Video; Perioperative Alleviation of Anxiety; Maternal Satisfaction; Preoperative Education; Elective Cesarean Section; Spinal Anesthesia
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The parturient will be randomly grouped into two groups which are Group V (Informative Video) and Group C (control group) using a computer-generated sequence in a permuted block of six. A research assistant/medical officer who is not involved in the conduct of study will perform the allocation concealment by placing the randomization sequence into sealed and opaque envelopes, which will be numbered accordingly. The next available envelope will be taken for the next recruited parturient and open by the investigator after the baseline anxiety level assessment is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group V ( Informative Video ) (Experimental): Receive QR code of the informative video. Participants can watch it on their phones as many times as they wish.
  During day of surgery , will receive standard care as per protocols .
  Interventions: Behavioral: Informative Video on Perioperative Anxiety and Maternal Satisfaction
- Group C ( Control Group ) (No Intervention): Will not receive the informative video . During day of surgery , will receive standard care as per protocols .

INTERVENTIONS:
Behavioral: Informative Video on Perioperative Anxiety and Maternal Satisfaction — An informative video designed to address potential sources of perioperative anxiety and dissatisfaction during elective lower segment caesarean section under spinal anaesthesia. The video provides details about the procedure, expected sensations, and management of discomfort to enhance patient understanding and reduce anxiety. It is administered to the intervention group of patients scheduled for elective caesarean section, allowing them to view it on their personal devices before the surgery.
  Arms: Group V ( Informative Video )

SUMMARY:
Title:

"Study of Informative Video on Alleviating Perioperative Anxiety and Improving Satisfaction Score in Obstetric Patients Undergoing Elective Lower Segment Caesarean Section Under Spinal Anaesthesia"

Objective:

This study aims to evaluate the effectiveness of an informative video in reducing perioperative anxiety and enhancing satisfaction in obstetric patients undergoing elective Caesarean sections under spinal anaesthesia. The hypothesis is that patients who view the video will experience lower anxiety and higher satisfaction compared to those who receive standard pre-anaesthetic counselling alone.

Background:

Spinal anaesthesia, commonly used for Caesarean sections, offers rapid, predictable pain relief but can cause discomfort due to factors such as visceral pain and fundal pressure, leading to perioperative anxiety. Anxiety can negatively impact maternal satisfaction and increase the risk of postpartum complications. Previous studies have shown mixed results regarding the efficacy of educational videos in alleviating this anxiety.

Methods:

The study is a prospective, randomized controlled trial conducted at Universiti Malaya Medical Centre. Eligible participants are obstetric patients (ASA II-III) undergoing elective Caesarean sections. Participants are randomly assigned to either an intervention group, which receives a supplemental informative video, or a control group receiving standard care. Anxiety and satisfaction levels are assessed using validated questionnaires pre- and post-surgery.

Anticipated Outcomes:

The study hypothesizes that the informative video will significantly reduce perioperative anxiety and improve maternal satisfaction, thereby demonstrating the superiority of this intervention over standard pre-anaesthetic counselling.

DETAILED DESCRIPTION:
Introduction Spinal anaesthesia is the preferred method for Caesarean sections due to its high success rate and minimal impact on maternal-fetal physiology. However, it is not without discomfort, as patients remain awake and can experience visceral pain, nausea, and other sensations that contribute to perioperative anxiety and dissatisfaction. This study explores the potential of an informative video to address these issues and improve patient outcomes.

Problem Statement Despite the widespread use of educational videos, the optimal approach for reducing anxiety and improving satisfaction in Caesarean patients remains unclear. Previous videos have focused on technical aspects of spinal anaesthesia without adequately addressing potential discomforts. This study seeks to bridge this gap by emphasizing specific sources of discomfort in the video content.

Research Questions Can an informative video highlighting potential sources of anxiety and dissatisfaction effectively alleviate these issues during the perioperative period? Is the video more effective than standard pre-anaesthetic counselling alone? Hypotheses Null Hypothesis: There is no significant difference in anxiety and satisfaction between patients who view the video and those who do not.

Alternative Hypothesis: Patients who view the video will have lower anxiety and higher satisfaction levels.

Objectives Evaluate if the video effectively reduces perioperative anxiety and dissatisfaction.

Determine if the video outperforms standard counselling in achieving these outcomes.

Methods

Study Design:

A prospective, randomized controlled trial at Universiti Malaya Medical Centre from July 2024 to June 2025.

Participants:

Inclusion Criteria: Obstetric patients ASA II-III undergoing first elective Caesarean section under spinal anaesthesia.

Exclusion Criteria: Patients under 18, ASA IV, diagnosed with morbid fetal conditions, or with psychiatric illness.

Randomization:

Participants are randomly assigned to two groups (Group V: Video, Group C: Control) using a computer-generated sequence. Allocation concealment is ensured through sealed envelopes.

Intervention:

The intervention group receives a QR code to access the informative video on their phones, with no viewing restrictions. The control group receives standard care.

Assessment Tools:

Anxiety: Spielberger State-Trait Anxiety Inventory (STAI), assessing pre- and post-operative anxiety levels.

Satisfaction: Maternal Satisfaction Scale for Caesarean Section (MSSCS), evaluating satisfaction post-surgery.

Sample Size:

A total of 75 participants (31 per group, accounting for a 20% dropout rate) are needed to detect a clinically significant reduction in anxiety.

Data Collection and Analysis Data are collected using standardized forms and questionnaires. Analysis is conducted with IBM SPSS to assess normal distribution and differences between groups. Statistical significance is determined at a p-value < 0.05.

Conclusion The study aims to demonstrate that an informative video addressing specific discomforts associated with spinal anaesthesia can significantly reduce anxiety and improve satisfaction in obstetric patients, offering a potentially superior alternative to standard pre-anaesthetic counselling.

ELIGIBILITY:
Inclusion Criteria:

* All obstetric patients American Society of Anaesthesiologists (ASA) II-III
* First time undergo elective caesarean section
* Under spinal anaesthesia.

Exclusion Criteria:

* Less than 18 years old
* ASA IV
* known antenatal diagnosis of morbid foetal conditions
* history of psychiatry illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Perioperative Anxiety Level | Preoperative: Baseline anxiety levels are assessed one day before the caesarean section.Postoperative: Anxiety levels are reassessed on day 1 post-caesarean section.
  The primary outcome measure is the level of perioperative anxiety experienced by patients, assessed using the Speiberger State-Trait Anxiety Inventory (STAI). This tool evaluates both state and trait anxiety levels, focusing on current anxiety experienced by patients before and after the elective lower segment caesarean section under spinal anaesthesia.

SECONDARY OUTCOMES:
Maternal Satisfaction with Anesthesia and Procedure | Postoperative: Maternal satisfaction is assessed on day 1 post-caesarean section, during the same time frame as the anxiety reassessment.
  The secondary outcome measure is maternal satisfaction, assessed using the Maternal Satisfaction Scale for Caesarean Section (MSSCS). This scale evaluates patients' overall satisfaction with their anaesthetic experience, including procedural comfort and management of any adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Kamarrudin Hadri, MBBS, Study Director — University of Malaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan YK, Ng KP. A survey of the current practice of obstetric anaesthesia and analgesia in Malaysia [correction of Malaysis]. J Obstet Gynaecol Res. 2000 Apr;26(2):137-40. doi: 10.1111/j.1447-0756.2000.tb01297.x. PMID 10870307
- [Result] Jiang A, Perry T, Walker K, Burfoot A, Patterson L. Surgical sensation during caesarean section: a qualitative analysis. Int J Obstet Anesth. 2024 Feb;57:103935. doi: 10.1016/j.ijoa.2023.103935. Epub 2023 Nov 3. PMID 37925355
- [Result] Vogel TM, Homitsky S. Antepartum and intrapartum risk factors and the impact of PTSD on mother and child. BJA Educ. 2020 Mar;20(3):89-95. doi: 10.1016/j.bjae.2019.11.005. Epub 2020 Jan 28. No abstract available. PMID 33456935
- [Result] Vogel H, Schaaf W, Jacob M. [Video-assisted patient education in anesthesia : How do medical users assess the procedure?]. Anaesthesist. 2018 Nov;67(11):829-836. doi: 10.1007/s00101-018-0496-4. Epub 2018 Oct 9. German. PMID 30302517
- [Result] Maghalian M, Mohammad-Alizadeh-Charandabi S, Ranjbar M, Alamdary FA, Mirghafourvand M. Informational video on preoperative anxiety and postoperative satisfaction prior to elective cesarean delivery: a systematic review and meta-analysis. BMC Psychol. 2024 Jan 2;12(1):6. doi: 10.1186/s40359-023-01499-3. PMID 38167236
- [Result] Lin SY, Huang HA, Lin SC, Huang YT, Wang KY, Shi HY. The effect of an anaesthetic patient information video on perioperative anxiety: A randomised study. Eur J Anaesthesiol. 2016 Feb;33(2):134-9. doi: 10.1097/EJA.0000000000000307. PMID 26196527
- [Result] Che YJ, Gao YL, Jing J, Kuang Y, Zhang M. Effects of an Informational Video About Anesthesia on Pre- and Post-Elective Cesarean Section Anxiety and Recovery: A Randomized Controlled Trial. Med Sci Monit. 2020 Apr 8;26:e920428. doi: 10.12659/MSM.920428. PMID 32265432
- [Result] Singh K, Heralal H. The Effect of a Simple Perioperative Video on Maternal Anxiety and Satisfaction Before Regional Anesthesia in a Caribbean Setting: A Randomized Controlled Trial. Cureus. 2023 Mar 21;15(3):e36482. doi: 10.7759/cureus.36482. eCollection 2023 Mar. PMID 37090355
- [Result] Abate, S. M., Chekol, Y. A., & Basu, B. (2020). Global prevalence and determinants of preoperative anxiety among surgical patients: A systematic review and meta-analysis. International Journal of Surgery Open, 25, 6-16
- [Result] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Result] Bansal T, Joon A. A comparative study to assess preoperative anxiety in obstetric patients undergoing elective or emergency cesarean section. Anaesth Pain Intensive Care 2019:25e30.
- [Result] Fentie Y, Yetneberk T, Gelaw M. Preoperative anxiety and its associated factors among women undergoing elective caesarean delivery: a cross-sectional study. BMC Pregnancy Childbirth. 2022 Aug 17;22(1):648. doi: 10.1186/s12884-022-04979-3. PMID 35978308
- [Result] Mitchell M. Conscious surgery: influence of the environment on patient anxiety. J Adv Nurs. 2008 Nov;64(3):261-71. doi: 10.1111/j.1365-2648.2008.04769.x. Epub 2008 Sep 10. PMID 18785887
- [Result] Matthey PW, Finegan BA, Finucane BT. The public's fears about and perceptions of regional anesthesia. Reg Anesth Pain Med. 2004 Mar-Apr;29(2):96-101. doi: 10.1016/j.rapm.2003.10.017. PMID 15029543
- [Result] Snyder-Ramos SA, Seintsch H, Bottiger BW, Motsch J, Martin E, Bauer M. Patient satisfaction and information gain after the preanesthetic visit: a comparison of face-to-face interview, brochure, and video. Anesth Analg. 2005 Jun;100(6):1753-1758. doi: 10.1213/01.ANE.0000153010.49776.E5. PMID 15920209
- [Result] Yılmaz, G., Akça, A., Esen, O., & Salihoğlu, Z. (2019). Multimedia education on the day of elective cesarean section increases anxiety scores. Perinatal Journal, 27(1), 38-42.
- [Result] Noben L, Goossens SMTA, Truijens SEM, van Berckel MMG, Perquin CW, Slooter GD, van Rooijen SJ. A Virtual Reality Video to Improve Information Provision and Reduce Anxiety Before Cesarean Delivery: Randomized Controlled Trial. JMIR Ment Health. 2019 Dec 18;6(12):e15872. doi: 10.2196/15872. PMID 31850850
- [Result] Kanyeki T, Mung'ayi V, Bal R, Odaba D. Effect of video-based information on preoperative State trait anxiety inventory scores in adult patients presenting for elective caesarean section: a randomized controlled trial. Afr Health Sci. 2022 Sep;22(3):117-124. doi: 10.4314/ahs.v22i3.14. PMID 36910414
- [Result] Eley VA, Searles T, Donovan K, Walters E. Effect of an anaesthesia information video on preoperative maternal anxiety and postoperative satisfaction in elective caesarean section: a prospective randomised trial. Anaesth Intensive Care. 2013 Nov;41(6):774-81. doi: 10.1177/0310057X1304100613. PMID 24180719
- [Result] Fisher PL, Durham RC. Recovery rates in generalized anxiety disorder following psychological therapy: an analysis of clinically significant change in the STAI-T across outcome studies since 1990. Psychol Med. 1999 Nov;29(6):1425-34. doi: 10.1017/s0033291799001336. PMID 10616949
- [Result] Spielberger C, Gorsuch R, Lushene R: State-trait anxiety inventory for adults sampler set: Manual, instrument and scoring guide. Consulting Psychologists Press, 1983
- [Result] Embong, H. (2018). Psychometric Properties of the Malay Translated Spielberger State-Trait Anxiety Inventory in Exploring Parental Anxiety. Medicine & Health, 13(1), 106-116.
- [Result] Morgan PJ, Halpern S, Lo J. The development of a maternal satisfaction scale for caesarean section. Int J Obstet Anesth. 1999 Jul;8(3):165-70. doi: 10.1016/s0959-289x(99)80132-0. PMID 15321139